CLINICAL TRIAL: NCT02779647
Title: Play as a Method to Reduce Overweight and Obesity in Children. Kids-Play Study.
Brief Title: Play as a Method to Reduce Overweight and Obesity in Children.
Acronym: Kids-Play
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, María José Aguilar Cordero, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01052013UGR
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Childhood Obesity; Sleep Apnea in Obese Children; Studying Maternal and Family Factors That Cause Obesity in Children
Keywords: Overweight, obesity, play, physical activity, accelerometry.
MeSH Terms: conditions — Pediatric Obesity; Overweight; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Experimental): Consisting of 49 children who were recommended a programme of physical activity, play and nutritional advice, for both the children and their parents
  Interventions: Behavioral: The intervention consisted of physical activity based on play
- Control group (No Intervention): 49 children, who received only nutritional advice

INTERVENTIONS:
Behavioral: The intervention consisted of physical activity based on play — The intervention consisted of physical activity based on play, with four 90-minute sessions per week for nine months (the school year). The total of sessions was 144, the minimum number of sessions to consider valid that a child has completed the intervention was 115 (80%) in order to perform the minimum level of physical activity recommended for their ages. In parallel, twice-monthly theoretical and practical sessions of nutritional advice were given to the children and their families. The study group performed the physical activity and received the nutritional advice, while the control group received only the theoretical and practical sessions on nutrition.
  Arms: Study group

SUMMARY:
Introduction Overweight and obesity are characterised by excess fat, which results in weight gain and is identified by the Body Mass Index (BMI). Studies show that overweight and obesity are the result of a complex interaction between genetic and environmental factors, which begins prenatally. Various studies have shown that physical exercise is an important component of weight loss programmes and that it also benefits the metabolic profile. Other authors have reported that greater weight loss is achieved by a programme that includes both diet and exercise, rather than either of these alone.

Aim The aim of this study is to analyse an intervention based on play as a means of improving the body composition of children with overweight or obesity.

Design / Method The design of the Kids-Play study is based on cases and controls. The study was conducted in Granada (Spain) The analysis sample of 98 children was divided into two groups: cases, consisting of 49 children, who participated in an intervention programme based on physical activity, play and nutritional advice (to both the child and the parents); and controls, another 49 children, who received only nutritional advice.

ELIGIBILITY:
Inclusion Criteria:

* Obese children that want participate in a voluntary way in the research and sign the informed consent.

Exclusion Criteria:

* Refused to participate
* Hormonal problems
* Age < 8 or >12 years
* Orthopaedic, respiratory
* Other problems

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Children's body composition | 12 months
  The children's body composition was measured before and after the intervention, by bioelectrical impedance and using the InBody 720 body composition analyser.

SECONDARY OUTCOMES:
The level of daily physical activity | 1 month
  The level of daily physical activity was assessed using ActiGraph wGT3X-BT accelerometers, which were worn on the right hip by all children in the study population for seven days, except during the hours of sleep. In this way it was possible to objectively analyse whether the study group met the WHO recommended levels of activity for their age group, and to determine the differences between cases and controls.
Sleep apnea | 6 month
  Sleep apnea has been measured by sleep polygraphy.

REFERENCES:
- [Derived] Sanchez-Lopez AM, Menor-Rodriguez MJ, Sanchez-Garcia JC, Aguilar-Cordero MJ. Play as a Method to Reduce Overweight and Obesity in Children: An RCT. Int J Environ Res Public Health. 2020 Jan 3;17(1):346. doi: 10.3390/ijerph17010346. PMID 31947884
- [Derived] Aguilar-Cordero MJ, Rodriguez-Blanque R, Leon-Rios X, Exposito Ruiz M, Garcia Garcia I, Sanchez-Lopez AM. Influence of Physical Activity on Blood Pressure in Children With Overweight/Obesity: A Randomized Clinical Trial. Am J Hypertens. 2020 Feb 22;33(2):131-136. doi: 10.1093/ajh/hpz174. PMID 31678988
- See also: Original research — http://scielo.isciii.es/pdf/nh/v27n4/42_original31.pdf
- See also: Systematic review — http://www.aulamedica.es/nh/pdf/7680.pdf
- Available data/document: Study Protocol — http://scielo.isciii.es/pdf/nh/v28n3/22original18.pdf
- Available data/document: Study Protocol — http://scielo.isciii.es/pdf/nh/v28n3/23original19.pdf